CLINICAL TRIAL: NCT02676518
Title: Anti-Müllerian Hormone and Its Association With Glucose Intolerance and Metabolic Syndrome in Women With Polycystic Ovary Syndrome
Brief Title: AMH, Glucose Intolerance and Metabolic Syndrome in PCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Porntip Sirayapiwat, Principal Investigator, Chulalongkorn University
Other Study IDs: 057/2015
Record Dates: First submitted 2015-08-19; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; Serum anti-Mullerian hormone; glucose intolerance; metabolic syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Glucose Intolerance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * Serum anti-mullerian hormone level
  * Blood test for 2-hours 75 gram glucose tolerance test
  * Blood tests for total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- polycystic ovary syndrome women: PCOS women diagnosed by Rotterdam criteria visiting the Gynecologic Unit at King Chulalongkorn Memorial Hospital and meet the inclusion criteria and no exclusion criteria of the study
  Interventions: Other: serum

INTERVENTIONS:
Other: serum — Serum for serum anti-Mullerian hormone, 2-hour 75 gram oral glucose tolerance test and lipid profiles

SUMMARY:
Association between serum anti-Mullerian hormone (AMH) level and prevalence of glucose intolerance and metabolic syndrome in women with polycystic ovary syndrome (PCOS)

DETAILED DESCRIPTION:
* To study the association between serum anti-Mullerian hormone (AMH) level and glucose intolerance and metabolic syndrome in women with polycystic ovary syndrome (PCOS).
* Glucose intolerance is detected by 2-hours 75 gram oral glucose tolerance test (OGTT).
* Metabolic syndrome is diagnosed by using the Harmonized criteria; the presence of any 3 of 5 following risk factors constitutes a diagnosis of metabolic syndrome.

  1. Elevated waist circumference (> 80 cm in Asian women)
  2. Elevated triglycerides (> 150 mg/dL)
  3. Reduced HDL-cholesterol (< 50 mg/dL)
  4. Elevated blood pressure )systolic > 130 and/or diastolic > 85 mmHg)
  5. Elevated fasting glucose ( > 100 mg/dL)
* Percentage of glucose intolerance and metabolic syndrome in PCOS women as well was any differences in parameters between PCOS patients with and without glucose intolerance and metabolic syndrome will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnosed by Rotterdam criteria 2003

Exclusion Criteria:

* Pregnancy
* Previous any hormonal uses in the last 3 months
* Previous hypoglycemic drugs or insulin-sensitising agents use in the last 3 months
* Previous chemotherapy, ovarian surgery, pelvic irradiation
* Menopause

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Thai women with PCOS diagnosed by Rotterdam criteria 2003 who visit at Gynecological Department, King Chulalongkorn Memorial Hospital, Bangkok,Thailand
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Differences between serum AMH level between PCOS women with and without glucose intolerance and metabolic syndrome | 6 months
  Any differences between mean of serum AMH levels in PCOS with and without glucose intolerance and metabolic syndrome

SECONDARY OUTCOMES:
Percentage of glucose intolerance in PCOS women | 6 months
  Percentage of glucose intolerance detected by 75 g OGTT in PCOS women
Percentage of metabolic syndrome in PCOS women | 6 months
  Percentage of metabolic syndrome defined by the Harmonized criteria in PCOS women

CONTACTS AND LOCATIONS:
Overall Officials: Dhirapong Charoenvidya, MD, Study Chair — Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Department of Obstetrics and Gynecology, Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes